CLINICAL TRIAL: NCT06471972
Title: Biomarkers After Out-of-hospital Cardiac Arrest- a STEPCARE Substudy
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: University of Helsinki (Other); The George Institute (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Medical Research Institute of New Zealand (Other)
Responsible Party: Sponsor
Other Study IDs: STEPCARE biomarker substudy
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Arrest
Keywords: Biomarkers; Brain injury
MeSH Terms: conditions — Heart Arrest; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and PAX-RNA will be collected. Blood will be sampled at 12, 24, 48 and 72 h after inclusion in STEPCARE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult out-of-hospital cardiac arrest patients in participating sites of the STEPCARE trial: Patients will not be randomized within the biomarker substudy, but are already randomised as participants within the STEPCARE trial to either of 3 interventions

SUMMARY:
A prospective multicenter biomarker study with adult patients treated on

intensive care units after out-of-hospital cardiac arrest. Patients will be recruited from specific sites participating in the Sedation, Temperature and Pressure After Cardiac Arrest and Resuscitation (STEPCARE) trial. (ClinicalTrials.gov ID NCT05564754).

Blood samples will be collected at 12, 24, 48, and 72 hours after randomization in selected sites, aliquoted and frozen on-site. After trial completion, samples will be stored in a central biobank. Sample analysis will be performed in batch after trial completion. Functional outcome will be assessed at 30 days and 6 months after cardiac arrest.

DETAILED DESCRIPTION:
A prospective multicenter biomarker study with adult patients treated on intensive care units after out-of-hospital cardiac arrest. Patients will be recruited from specific sites participating in the Sedation, Temperature and Pressure After Cardiac Arrest and Resuscitation (STEPCARE) trial. (ClinicalTrials.gov ID NCT05564754). The STEPCARE-trial is a 2x2x2 randomised trial studying patients who have been resuscitated from cardiac arrest and who are comatose. It will include three different interventions focusing on sedation targets, temperature targets and mean arterial pressure targets.

3500 patients who are comatose after cardiac arrest will be included in the STEPCARE trial studying three separate targets. All patients will be randomised to a control or an intervention arm for sedation, temperature and blood pressure targets as follows:

* Continuous deep sedation for 36 hours or minimal sedation (SEDCARE)
* Fever management with or without a feedback-controlled device (TEMPCARE)
* A mean arterial pressure target of >85mmHg or >65mmHg. (MAPCARE)

Hospitals participating in the STEPCARE trial may opt to participate in the biomarker substudy if they include >20 patients/year, have the possibility to collect and process samples 24/7. Processing should be done by professional or experienced personnel.

Blood samples will be collected at 12, 24, 48, and 72 hours after randomization in selected sites, aliquoted and frozen on-site. Serum, plasma and PAX-RNA vials are collected. After trial completion, samples will be stored in a central biobank. Sample analysis will be performed in batch after trial completion.

Functional outcome will be assessed at 30 days and 6 months after cardiac arrest. Primary outcome is poor functional outcome (modified Rankin Scale 4-6) at six months. Secondary outcomes are poor functional outcome at 30 days and survival at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* From sites participating in the STEPCARE biomarker substudy and withOut-of-hospital cardiac arrest
* Sustained ROSC - defined as 20 minutes with signs of circulation without the need for chest compressions
* Unconsciousness defined as not being able to obey verbal commands (FOUR-score motor response of <4) or being intubated and sedated because of agitation after sustained ROSC.
* Eligible for intensive care without restrictions or limitations
* Inclusion within 4 hours of ROSC

Exclusion Criteria:

* On ECMO prior to randomization
* Pregnancy
* Suspected or confirmed intracranial hemorrhage
* Previously randomized in the STEPCARE trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an out-of-hospital cardiac arrest from sites participating in the biobank substudy of the STEPCARE trial will be included.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome according to the modified Rankin Scale | 6 months after randomisation
  Poor functional outcome modified Rankin Scale 4-6 (moderately severe disability, severe disability or death). A higher score indicates a worse score.

SECONDARY OUTCOMES:
Functional outcome according to the modified Rankin Scale | 30 days after randomisation
  Poor functional outcome modified Rankin Scale 4-6 (moderately severe disability, severe disability or death). A higher score indicates a worse score.
Mortality at 6 months | 6 months after randomisation
  Mortality from any cause at six months follow-up

CONTACTS AND LOCATIONS:
Locations (4):
- Helsinki Hospital, Helsinki, Finland
- Sweden (3):
  - Helsingborgs Hospital, Helsingborg
  - Skåne university hospital, Lund
  - Skåne University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request following publication.

REFERENCES:
- See also: Website for the trial — http://www.stepcare.org
- Available data/document: Study Protocol — http://stepcare.org/biomarkers — Lab manuals and sample collection form